CLINICAL TRIAL: NCT00562328
Title: Antibody Therapy With Alemtuzumab, Rituximab and GM-CSF for Initial Treatment of High Risk Chronic Lymphocytic Leukemia
Brief Title: Rituximab, Alemtuzumab, and GM-CSF As First-Line Therapy in Treating Patients With Early-Stage Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574754; P30CA015083 (NIH); MC0785 (Other: Mayo Clinic Cancer Center); U4449s (Other: Genentech); 001.0888 (Other: Bayer); 07-002087 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (1):
- Alemtuzumab + Rituximab + GM-CSF (Experimental): Alemtuzumab + Rituximab + GM-CSF
  Interventions: Biological: Alemtuzumab; Biological: Rituximab; Biological: Sargramostim

INTERVENTIONS:
Biological: Alemtuzumab — Week 1 (dose escalation):
  Day 3: 3mg subcutaneously; Day 4: 10mg subcutaneously; Day 5 30mg subcutaneously
  Weeks 2-5:
  30mg subcutaneously three times a week.
Biological: Rituximab — Weeks 2-5:
  375 mg/m^2 by IV once weekly
Biological: Sargramostim — Week 1-6:
  250 mcg subcutaneously three time as week
  Other Names: GM-CSF

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab and alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving monoclonal antibody therapy together with GM-CSF may be an effective treatment for early-stage chronic lymphocytic leukemia.

PURPOSE: This phase II trial is studying the side effects of giving rituximab and alemtuzumab together with GM-CSF and to see how well it works in treating patients with early-stage chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the rate of complete and overall response in patients with high-risk, early-stage, chronic lymphocytic leukemia (CLL) treated with alemtuzumab, rituximab, and sargramostim (GM-CSF).
* To monitor and assess toxicity of this regimen in these patients through clinical evaluation and serial monitoring of cytomegalovirus antigenemia by polymerase chain reaction (PCR).

Secondary

* To determine the overall and progression-free survival, time to response, time to next treatment, and duration of response in patients treated with this regimen.
* To assess the correlation between individual prognostic markers (i.e., 17p-, 11q-, unmutated VH gene, use of VH3-21, ZAP70+, CD38+) and clinical outcome.

Correlative Studies

* To assess response in these patients using an expanded definition of response, including minimal residual disease (MRD) by sensitive flow cytometry in patients in complete clinical remission.
* To assess MRD status of responding patients using sensitive flow cytometry and molecular assays (i.e., spectral karyotype analysis of CLL cells) before treatment and at relapse to identify subpopulations that could contribute to disease resistance and relapse.
* To detail the in vivo effect of this regimen on critical aspects of the immune system in CLL.
* To determine if GM-CSF, β-glucan, and CpG7909 can increase antibody dependent cellular cytotoxicity to improve efficacy against CLL cells and clinical response to treatment.

OUTLINE: Patients receive rituximab IV over 30 minutes on day 3 of weeks 2-5, alemtuzumab subcutaneously (SC) on days 3, 4, and 5 in week 1 and on days 1, 3, and 5 in weeks 2-5, and sargramostim SC on days 1, 3, and 5 in weeks 1-6. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection for measurement of serum cytomegalovirus DNA copy number by polymerase chain reaction at baseline, weekly during treatment, and monthly for the 6 months after completion of treatment. Patients also undergo bone marrow biopsy and aspirate at two months and then again at 12 months (if in complete remission). Blood samples are collected periodically during study for evaluation of prognostic biomarkers (i.e., 11q-, 17p-, unmutated IgVH gene, VH3-21 gene segment use, and CD38 and ZAP-70 expression) by fluorescent in situ hybridization (FISH) and for immunophenotyping by flow cytometry. Blood samples are collected from patients at the Mayo Clinic Rochester site at baseline and periodically during study for immunological and other correlative studies, including minimal residual disease (in responding patients only).

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) meeting the following criteria:

  * Minimum threshold peripheral blood lymphocyte count 5 x 10^9/L
  * Monoclonality (light chain exclusion) of B lymphocytes detected by immunophenotyping (CD19-positive), demonstrating ≥ 3 of the following characteristics:

    * CD5-positive
    * CD23-positive
    * Dim surface light chain expression
    * Dim surface CD20 expression
  * Negative for IGH/CCND1 translocation AND/OR immunostaining is negative for cyclin D1 expression by fluorescent in-situ hybridization (FISH) analysis
  * Rai stage 0, I, or II disease that does not meet standard NCI-Working Group criteria for treatment of CLL
* Poor prognosis as defined by ≥ 1 of the following factors:

  * Unmutated IgVH mutation status AND CD38 expression (i.e., ≥ 30% cells positive on flow cytometry)
  * Unmutated IgVH mutation status AND ZAP-70 expression (i.e., ≥ 20% cells positive on flow cytometry)
  * VH3-21 gene segment use irrespective of mutation status AND CD38 expression (≥ 30% cells positive on flow cytometry)
  * VH3-21 gene segment use irrespective of mutation status AND ZAP-70 expression (≥ 20% cells positive on flow cytometry)
  * 11q-negative*
  * 17p-negative* NOTE: *Determination of IgVH mutation status is not required in patients whose eligibility is based on 17p13- or 11q22- deletions

PATIENT CHARACTERISTICS:

* ECOG performance status 0- 2
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 3.0 times ULN OR direct bilirubin ≤ 1.5 ULN
* AST ≤ 3.0 times ULN (unless due to hemolysis or CLL)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must practice effective contraception
* Willing to provide mandatory blood samples (for patients at the Mayo Clinic in Rochester only) for research studies as required by the protocol
* No comorbid conditions, including any of the following:

  * New York Heart Association Class III or IV heart disease
  * Myocardial infarction within the past month
  * Uncontrolled infection
  * HIV infection or AIDS
  * Serological evidence of active hepatitis B infection (i.e., serum antigen or e-antigen positivity) or positive hepatitis C serology
* No other active primary malignancy requiring treatment or limiting survival to ≤ 2 years
* No active autoimmune hemolytic anemia, immune thrombocytopenia, or pure red blood cell aplasia

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior major surgery
* No prior chemotherapy or monoclonal antibody treatment for CLL
* No concurrent corticosteroids

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2010-02-05 (Actual); Study Completion 2014-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clive S. Zent, MD, Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Derived] Zent CS, Wu W, Bowen DA, Hanson CA, Pettinger AM, Shanafelt TD, Kay NE, Leis JF, Call TG. Addition of granulocyte macrophage colony stimulating factor does not improve response to early treatment of high-risk chronic lymphocytic leukemia with alemtuzumab and rituximab. Leuk Lymphoma. 2013 Mar;54(3):476-82. doi: 10.3109/10428194.2012.717276. Epub 2012 Aug 22. PMID 22853816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-three (33) participants were recruited at Mayo Clinic (Rochester and Arizona) between January 2008 and February 2010.
Pre-assignment Details: All patients were deemed eligible.
Period: Overall Study
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 60 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 33
Rai Stage [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity.
  Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis and lymphadenopathy, Rai Stage II: Lymphocytosis and hepatomegaly +/- splenomegaly, Rai Stage III: Lymphocytosis and anemia, Rai Stage IV: Lymphocytosis and thrombocytopenia
  participants
    Stage 0 | 2
    Stage 1 | 27
    Stage 2 | 4
CD38 Expression Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive CD38 (>=30%) tend to experience a more aggressive course of CLL.
  participants
    Positive (>=30%) | 15
    Negative (<30%) | 18
Immunoglobulin Variable Heavy Chain (IGVH) Mutation Status [Number; unit: participants] — IGVH testing helps predict which patients will experience a more aggressive (if the gene is unmutated, <=2%) or less aggressive (if the gene is mutated, >2%) course of CLL. This technically complex test is only available at select medical institutions.
  participants
    Mutated | 3
    Unmutated | 30
ZAP-70 Expression [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive ZAP-70 (>=20%) tend to experience a more aggressive course of CLL.
  participants
    Positive (>=20%) | 25
    Negative (<20%) | 7
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Confirmed Responses (Complete or Partial Response Noted as the Objective Status for a Duration of at Least 2 Months) at 6 Months
Description: Response, as defined by the National Cancer Institute Working Group (NCIWG), requires the following for a period of at least 2 months:
  * CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy
  * PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100,000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Alemtuzumab + Rituximab + GM-CSF: Patients received Alemtuzumab + Rituximab + GM-CSF.
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Number analyzed (Participants) | 33
Participants | 31

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to the standard NCI-WG96 criteria. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from registration to progression (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Number analyzed (Participants) | 33
months | 13.0 [9.4 to NA] — The 95% confidence interval upper limit was not yet reached (below the level of detection).

3. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) is defined as the time from documentation of response (CR or PR) to disease progression. The median DOR with 95% CI was estimated using the Kaplan Meier method.Response, as defined by the National Cancer Institute Working Group (NCIWG), requires the following for a period of at least 2 months:
  * CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy
  * PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100,000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions
Time Frame: time from start of response to progression (up to 5 years)
Population: Only patients who responded to treatment are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Number analyzed (Participants) | 31
months | 14.9 [8.8 to NA] — The 95% confidence interval upper limit was not yet reached (below the level of detection).

4. Secondary Outcome: Time to Next Treatment
Description: Time to next treatment was defined as the time from end of active (protocol) treatment to the start of subsequent treatment. The median and 95% CI was estimated using the Kaplan Meier method.
Time Frame: time from end of protocol treatment to subsequent treatment (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Number analyzed (Participants) | 33
months | 33.5 [25.5 to NA] — The 95% confidence interval upper limit was not yet reached (below the level of detection).

5. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from registration to death of any cause. Participants were followed for a maximum of 5 years from registration. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Time from registration to death (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Number analyzed (Participants) | 33
months | NA [NA to NA] — Median and 95% confidence interval for overall survival has not been reached (below the level of detection).

ADVERSE EVENTS:
Arm/Group | Alemtuzumab + Rituximab + GM-CSF
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab + Rituximab + GM-CSF (N=33)
Pneumonia (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab + Rituximab + GM-CSF (N=33)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 3 (4)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 24 (43)
Injection site reaction (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Blood Infection (Infections and infestations) | 3 (5)
Bronchial infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (5)
Lip infection (Infections and infestations) | 1 (1)
Opportunisitic infection (Infections and infestations) | 3 (6)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 6 (9)
Bilirubin (Investigations) | 1 (3)
Leukopenia (Investigations) | 16 (39)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 7 (17)
Platelet count decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatology (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 25 (59)
Sweating (Skin and subcutaneous tissue disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes